CLINICAL TRIAL: NCT07206472
Title: A Multi-national, Non-interventional Study of Bempedoic Acid or Its Single-pill Combination Therapy With Ezetimibe in Routine Clinical Practice in Patients With Primary Hypercholesterolaemia or Mixed Dyslipidaemia
Brief Title: A Study of Bempedoic Acid or Its Single-pill Combination Therapy With Ezetimibe in Patients With Primary Hypercholesterolaemia or Mixed Dyslipidaemia
Acronym: Musashi
Status: Not yet recruiting | Type: Observational
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Other Study IDs: DS-ASCAHQ-BMP-HC001
Record Dates: First submitted 2025-09-25; First posted 2025-10-03 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Primary Hypercholesterolaemia; Mixed Dyslipidemia
Keywords: Primary hypercholesterolemia; Mixed dyslipidemia
MeSH Terms: interventions — Ezetimibe

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Bempedoic acid/FDC with ezetimibe: Adult participants who were diagnosed with primary hypercholesterolemia (heterozygous familial and nonfamilial) or mixed dyslipidemia and treated with bempedoic acid/fixed dose combination (FDC) with ezetimibe in a regular clinical care setting.
  Interventions: Drug: Combination of bempedoic acid and ezetimibe

INTERVENTIONS:
Drug: Combination of bempedoic acid and ezetimibe — No drug was administered in this observational study.

SUMMARY:
There is limited efficacy and safety data of bempedoic acid or its fixed dose combination (FDC) with ezetimibe in Asian and Latin American patients. This non-interventional study (NIS) will be conducted to characterize the risks and benefits of bempedoic acid or FDC with ezetimibe in a real-world clinical setting in adult patients with primary hypercholesterolaemia (heterozygous familial and non-familial) or mixed dyslipidaemia.

DETAILED DESCRIPTION:
The primary objective of this study is to describe patient characteristics and evaluate adverse drug reactions (ADRs) that occurred since initiation of bempedoic acid/FDC with ezetimibe and adverse events (AEs) collected after signed informed consent and initiation of bempedoic acid/FDC with ezetimibe in a regular clinical care setting in patients with primary hypercholesterolaemia (heterozygous familial and non-familial) or mixed dyslipidaemia during 1-year follow-up.

The secondary objectives are defined as the assessment of the cardiovascular risk, rate, level of LDL-C goal attainment, changes over time in LDL-C levels, inflammatory markers, and uric acid levels from prior to treatment with bempedoic acid/FDC, and adverse events (AEs)/adverse drug reactions (ADRs).

ELIGIBILITY:
Patients can be enrolled, when they fulfil the following inclusion criteria:

* Written informed consent to participate.
* At least 18 years of age.
* Patients suffering from documented primary hypercholesterolemia or mixed dyslipidaemia treated or intended to be treated with bempedoic acid/ FDC with ezetimibe at the discretion of the physician are appropriate for participation in the observation.
* For patients who are treated with bempedoic acid/FDC with ezetimibe prior to signed informed consent, initiation of bempedoic acid/FDC with ezetimibe must be within a maximum of three months prior to inclusion.
* No contraindications exist according to the SmPC of bempedoic acid/FDC with ezetimibe.
* No concurrent participation in an interventional study (simultaneous participation in other non-interventional study is possible)
* Life expectancy > 1 year.

No explicit exclusion criteria exist to avoid selection bias and to allow for documentation of routine clinical practice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes adult patients diagnosed with primary hypercholesterolemia or mixed dyslipidemia treated by specialized as well as non-specialized physicians in hospitals and office-based centers from six countries (Brazil, Hong Kong, South Korea, Taiwan, Thailand, and Vietnam).
Sampling Method: Non-Probability Sample
Enrollment: 2560 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2028-09-01 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | From pre-bempedoic acid/pre-FDC initiation to 1 year after initiation of therapy
  Adverse events (AEs) will be collected after signed informed consent and initiation of bempedoic acid/FDC with ezetimibe.

SECONDARY OUTCOMES:
Cardiovascular (CV) risk of patients treated with bempedoic acid/FDC with ezetimibe using 2019 ESC/EAS guidelines risk classification | From pre-bempedoic acid/pre-FDC initiation to 1 year after initiation of therapy
  Cardiovascular (CV) risk of patients treated with bempedoic acid/FDC with ezetimibe will be assessed using 2019 ESC/EAS guidelines risk classification.
Proportion of patients with level of LDL-C goal attainment | From pre-bempedoic acid/pre-FDC initiation to 1 year after initiation of therapy
  The proportion of patients with level of LDL-C goal attainment at any subsequent data collection time point will be assessed.
Change from baseline in LDL-C levels | From pre-bempedoic acid/pre-FDC initiation to 1 year after initiation of therapy
  Changes over time in LDL-C levels from prior to treatment with bempedoic acid/FDC to any subsequent data collection points will be assessed.
Change from baseline in plasma levels of other potentially ASCVD-modifying cholesterol fragments | From pre-bempedoic acid/pre-FDC initiation to 1 year after initiation of therapy
  Changes over time in plasma levels of other potentially atherosclerotic cardiovascular disease (ASCVD)-modifying cholesterol fragments, namely, TC, apoB, HDL-C, non-HDL-C, TGs and Lp(a) from prior to treatment with bempedoic acid/FDC with ezetimibe to any subsequent data collection point will be assessed.
Change from baseline in the levels of inflammatory marker hsCRP | From pre-bempedoic acid/pre-FDC initiation to 1 year after initiation of therapy
  Changes over time in the levels of inflammatory marker Hs C-reactive Protein (hsCRP) from prior to treatment with bempedoic acid/FDC with ezetimibe to any subsequent data collection point will be assessed.
Change from baseline in uric acid levels | From pre-bempedoic acid/pre-FDC initiation to 1 year after initiation of therapy
  Changes over time in uric acid levels from prior to treatment with bempedoic acid/FDC with ezetimibe to any subsequent data collection point will be assessed.
Incidence of relevant cardiovascular events | From pre-bempedoic acid/pre-FDC initiation to 1 year after initiation of therapy
  The incidence of relevant CV events, including myocardial infarction (MI), unstable angina requiring hospitalization, CABG, PCI, stroke (ischemic and haemorrhagic), TIA , acute peripheral arterial occlusion, other arterial revascularization procedures, all-cause death, and CV-death will be assessed.
Adverse effects related to lipid-modifying treatments (LMTs) other than bempedoic acid/FDC with ezetimibe | From pre-bempedoic acid/pre-FDC initiation to 1 year after initiation of therapy
  Adverse effects related to lipid-modifying treatment (LMT) other than bempedoic acid/FDC with ezetimibe, including insufficient lipid lowering efficacy, laboratory abnormalities, muscle-associated symptoms, new onset and/or worsening of existing diabetes mellitus, reduced kidney function, drug-drug interaction assessed by the physician, and non-compliance assessed by the physician will be assessed.
Use of lipid modifying therapies prior or concomitantly to receiving bempedoic acid/FDC with ezetimibe | From pre-bempedoic acid/pre-FDC initiation to 1 year after initiation of therapy
  The use of LMTs prior or concomitantly to receiving bempedoic acid/FDC with ezetimibe (including combination treatments) will be assessed.
Treatment duration of bempedoic acid/FDC with ezetimibe | From pre-bempedoic acid/pre-FDC initiation to 1 year after initiation of therapy
  Bempedoic acid/FDC with ezetimibe treatment parameters such as treatment duration by therapy, dosage, prescription intervals, permanent discontinuations, switches and reasons for these will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Global Team Lead, Study Director — Daiichi Sankyo

IPD SHARING:
Plan to Share IPD: No